CLINICAL TRIAL: NCT04415892
Title: The Role of Transient Receptor Potential Channels in Chemotherapy-Induced Peripheral Neuropathic Pain.
Brief Title: The Role of TRP Channels in CIPN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CCP19-3307-CIPN
Record Dates: First submitted 2020-05-20; First posted 2020-06-04 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-02

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Cinnamaldehyde; Capsaicin; Dermal Blood Flow; Fingers; Human; Reproducibility; Paclitaxel; Oxaliplatin; Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — cinnamaldehyde; Capsaicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Healthy volunteers (Other): Young, healthy male volunteers to characterize the DBF changes upon cinnamaldehyde and capsaicin, including the reproducibility.
  Interventions: Other: Cinnamaldehyde and capsaicin
- Paclitaxel Patients (Other): Group of patients after treatment with paclitaxel.
  Interventions: Other: Cinnamaldehyde and capsaicin
- Paclitaxel Controls (Other): Group of healthy volunteers, matched for sex, age and BMI with the group of Paclitaxel Patients.
  Interventions: Other: Cinnamaldehyde and capsaicin
- Oxaliplatin Patients (Other): Group of patients after treatment with oxaliplatin.
  Interventions: Other: Cinnamaldehyde and capsaicin
- Oxaliplatin Controls (Other): Group of healthy volunteers, matched for sex, age and BMI with the group of Oxaliplatin Patients.
  Interventions: Other: Cinnamaldehyde and capsaicin
- Longitudinal Paclitaxel Patients (Other): Group of patients who are treated with paclitaxel.
  Interventions: Other: Cinnamaldehyde and capsaicin
- Longitudinal Oxaliplatin Patients (Other): Group of patients who are treated with oxaliplatin.
  Interventions: Other: Cinnamaldehyde and capsaicin

INTERVENTIONS:
Other: Cinnamaldehyde and capsaicin — Topical application of cinnamaldehyde and capsaicin on the fingers

SUMMARY:
Part I:

Evaluating the increase in dermal blood flow upon topical application of cinnamaldehyde and capsaicin on the fingers in healthy, male volunteers. In addition, the inter-period and inter-hand reproducibility of the increase in dermal blood flow will be assessed.

Part II:

Evaluating the increase in dermal blood flow upon topical application of cinnamaldehyde and capsaicin on the fingers in patients suffering from chemotherapy-induced peripheral neuropathy compared to matched healthy volunteers.

Part III:

Evaluating the increase in dermal blood flow upon topical application of cinnamaldehyde and capsaicin on the fingers in patients who are treated with paclitaxel or oxaliplatin.

DETAILED DESCRIPTION:
The primary aim is to investigate whether paclitaxel and/or oxaliplatin alter TRP channel functionality in vivo in human. TRP functionality can indirectly be assessed via dermal blood flow changes which are part of the so-called neurogenic inflammation, induced upon TRP activation. In vivo in human, TRP can be activated via topical application of cinnamaldehyde or capsaicin on the skin.

In Part I of the study, the DBF changes upon topical application of cinnamaldehyde or capsaicin on the fingers will be characterized, including inter-period and inter-hand reproducibility.

In Part II, patients who are suffering from chronic CIPN after treatment with paclitaxel or oxaliplatin are included. DBF changes upon cinnamaldehyde and capsaicin are compared to a matched control group.

In Part III, DBF changes are assessed in patients prior to the first administration of taxol/oxaliplatin and at regular points in time during the dosage regimen.

ELIGIBILITY:
Inclusion Criteria Healthy volunteers:

1. Subject is a white male ≥18 and ≤45 years of age.
2. Subject is a non-smoker for at least 6 months prior to the start of the study.
3. Subject has a body mass index between 18-30 kg/m².
4. Subject is judged to be in good health on the basis of medical history, physical examination and vital signs.
5. Subject understands the procedures and agrees to participate in the study by giving written informed consent.
6. Subject is matched to the patient groups for sex, age and BMI (only part II).

Inclusion Criteria Patients of Part II:

1. Subject is a white male or female ≥18 and ≤70 years of age.
2. Subject is a non-smoker for at least 6 months prior to the start of the study.
3. Subject has a BMI between 18-35 kg/m².
4. Subject has a history of treatment with one of the following chemotherapeutic agents:

   * Paclitaxel
   * Oxaliplatin
5. Subject suffers from peripheral neuropathy grade 1, 2 or 3 according to the Total Neuropathy Score (clinical version). Grade 1 correlates to a score of 1-7, grade 2 to a score of 8-14 and grade 3 to a score of 15-21(10-12).
6. Subject suffers from neuropathic symptoms in the upper limbs.
7. Discontinuation or termination of therapy with the chemotherapeutic agent occurred >1 month and < 1 year ago.
8. Subject understands the procedures and agrees to participate in the study by giving written informed consent.

Inclusion Criteria for patients of Part III

1. Subject is a white male or female ≥18 and ≤75 years of age.
2. Subject is a non-smoker for at least 6 months prior to the start of the study.
3. Subject has a BMI between 18-35 kg/m².
4. Subject will receive treatment with paclitaxel or oxaliplatin in the near future.
5. Subject understands the procedures and agrees to participate in the study by giving written informed consent.

Exclusion Criteria:

1. Subject has eczema, scleroderma, psoriasis, dermatitis, or keloids, tumors, ulcers, burns, flaps or grafts on their fingers or any other abnormality of the skin which, in the opinion of the investigator may interfere with the study assessments.
2. Subject has excessive hair growth on the fingers.
3. Subject cannot avoid excessive tanning (any exposure to sunlight or a tanning bed which would cause a sunburn reaction) throughout the study.
4. Subject has a history of significant severe (drug) allergies.
5. Subject uses any prescription or non-prescription drugs on a regular basis which, in the investigator's opinion, might confound the results of the study.
6. Subject currently uses lotions, oils, depilatory preparations, makeup, or other topical treatments on the fingers on a regular basis which cannot be discontinued for the duration of the study.
7. Subject is unable to refrain from drinking alcohol 24 hours prior to each study visit, is currently a regular user of any illicit drugs, or has a history of drug (including alcohol) abuse.
8. Subject is unable to refrain from drinking caffeinated beverages (e.g. coffee, tea, cola, …) 24 hours prior to each study visit. Subject is unable to limit their intake of caffeinated beverages to ≤4 cups a day throughout the study.
9. Subject has any of the following vital sign measurements at screening after at least 10 minutes of supine rest: Heart Rate <40 or >100 beats/min, Diastolic Blood Pressure <50 or >90 mmHg, Systolic Blood Pressure <90 or >140 mmHg.
10. Subject is currently participating or has been involved in testing an investigational drug in another clinical study within the last 4 weeks.
11. Subject is in a situation or has a condition which, in the opinion of the investigator, may interfere with safe and optimal participation in the study.
12. Subject has a history of any illness or disorder which, in the investigator's opinion, might confound the results of the study.
13. Subject suffered from peripheral neuropathy prior to the chemotherapeutic treatment (Only for patients).
14. Subject has (a history of) diabetes mellitus, amyloidosis, vitamin B deficiency or any other medical disorder that, in the investigator's opinion, may cause peripheral neuropathy (only for Part II and III).
15. Subject has (a history of) a lesion in the central nervous system that is known to possibly cause neuropathic pain: e.g. spinal cord injury, infarction localized in the brainstem or thalamus, syringomyelia, multiple sclerosis, or any other disorder of the CNS that, in the investigator's opinion, may cause neuropathic pain (only for Part II and III).
16. Subject has a history of treatment with bortezomib, vincristine, or any other compound that, in the investigator's opinion, may cause neuropathic pain (only for Part II and III).
17. Subject did not develop neuropathy after treatment with epirubicine-cyclofosfamide (only for the paclitaxel group in Part III).
18. Subject has a family history of peripheral neuropathy (only for Part II and III).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Characterization cinnamaldehyde | Dermal blood flow response measured during 60 minutes post-application
  The dermal blood flow response to topical application of cinnamaldehyde as assessed by LASCA on the fingers in healthy, male volunteers.
Inter-hand reproducibility cinnamaldehyde | Dermal blood flow response measured simultaneously on both hands during 60 minutes post-application during study visit 1
  The within subject inter-hand reproducibility of the dermal blood flow response to topical application of cinnamaldehyde as assessed by LASCA on the fingers in healthy, male volunteers
Inter-period reproducibility cinnamaldehyde | Interval of at least 5 days between both periods
  The within subject inter-period reproducibility (i.e. assessing changes) of the dermal blood flow response to topical application of cinnamaldehyde as assessed by LASCA on the fingers in healthy, male volunteers
Characterization capsaicin | Dermal blood flow response measured during 60 minutes post-application
  The dermal blood flow response to topical application of capsaicin as assessed by LASCA on the fingers in healthy, male volunteers
Inter-hand reproducibility capsaicin | Dermal blood flow response measured simultaneously on both hands during 60 minutes post-application during study visit 3
  The within subject inter-hand reproducibility of the dermal blood flow response to topical application of capsaicin as assessed by LASCA on the fingers in healthy, male volunteers.
Inter-period reproducibility capsaicin | Interval of at least 5 days between both periods
  The within subject inter-period reproducibility (i.e. assessing changes) of the dermal blood flow response to topical application of capsaicin as assessed by LASCA on the fingers in healthy, male volunteers.
DBF patients compared to healthy volunteers | Dermal blood flow measured in patients who are suffering from CIPN 1 to 12 months after the last administration of paclitaxel or oxaliplatin.
  The dermal blood flow changes upon topical application of cinnamaldehyde and capsaicin in patients suffering from chemotherapy-induced peripheral neuropathy compared to matched healthy volunteers.
DBF in patients before, during and after chemotherapeutic treatment | Dermal blood flow measured prior to the first, or within 5 days after administration of paclitaxel or oxaliplatin
  The dermal blood flow changes upon topical application of cinnamaldehyde and capsaicin in patients prior to, during and after treatment with either paclitaxel or oxaliplatin.

CONTACTS AND LOCATIONS:
Overall Officials: Jan de Hoon, MD, PhD, MSc, Principal Investigator — Center for Clinical Pharmacology
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No